CLINICAL TRIAL: NCT03638492
Title: Long-term Follow-up of Survival in Surgical Resected Invasive Cutaneous Melanomas: Comparing 2-cm Versus 4 -cm Resection Margins - a Randomized, Multicenter Trial
Brief Title: Trial of Surgical Excision Margins in Thick Primary Melanoma - 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peter Gillgren (Other)
Responsible Party: Sponsor-Investigator, Peter Gillgren, Head of Section for Vascular Surgery, Karolinska Institutet
Organization: Karolinska Institutet (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Margins Melanoma -2; Country specific (Other: Swe; Nat Reg Nr, Dk; 5 dig ser nr (8XXXX), Ea; 5 dig ser nr (7XXXX), Ny; 4 dig ser nr (9XXX))
Record Dates: First submitted 2018-08-07; First posted 2018-08-20 (Actual); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: Melanoma; Surgery; Treatment Outcome
Keywords: Melanoma/mortality/pathology/*surgery; Randomized Controlled Trials as Topic; Survival; Margin
MeSH Terms: conditions — Melanoma; Margins of Excision

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 cm margin of excision (Active Comparator): Patients with CMM >2 mm treated with an excision of 2-cm.
  Interventions: Procedure: 2-cm margin
- 4 cm margin of excision (Active Comparator): Patients with CMM >2 mm treated with an excision of 4-cm.
  Interventions: Procedure: 4-cm margin

INTERVENTIONS:
Procedure: 2-cm margin — Patients with CMM treated with a surgical safety margin of 2-cm in the surrounding skin and down to the fascia.
  Arms: 2 cm margin of excision
Procedure: 4-cm margin — Patients with CMM treated with a surgical safety margin of 4-cm in the surrounding skin and down to the fascia.
  Arms: 4 cm margin of excision

SUMMARY:
Objectives: The purpose of this study was to assess the long-term follow-up of the overall and melanoma-specific survival in the randomised, open-lable multicenter trial (NTC NCT01183936) comparing excision margin of 2 cm versus 4 cm for patients with primary cutaneous malignant melanoma (CMM) thicker than 2 mm.

Study hypothesis: The hypothesis is that there is no difference between the two treatment arms measured as melanoma-specific survival and overall survival.

DETAILED DESCRIPTION:
Historically, CMMs have been excised with wide resection margins of 5-cm or more with the radical removal of lymph nodes. This treatment emerged from a recommendation from Handley in 1907 based on a single pathological specimen. This "radical" surgical management resulted in bad cosmetic results, lymphedema, long hospital inpatient stay, frequent skin grafting and/or complicated skin flap reconstructions. Not until some 60-plus years later did questions arise in clinical practices whether the need for this extensive surgery was mandated and clinical practice was not substantially changed until the late 1980's. Retrospective studies published in the 1980s suggested that narrower excision margins may be appropriate for treatment of some CMMs, especially thinner lesions.

Nowadays, the recommendations for surgical treatment are based on the Breslow thickness of the CMM, since it is considered the most important prognostic indicator of localized disease and is therefore the information upon which today's surgical strategies are founded. However, recommendations vary over the world, especially for thicker tumors which is clearly presented by Ethun et al. (2016). For CMM of ≤ 1 mm thickness most centers use a 1 cm margin, but for tumors 1.01 - 4 mm the margins of resection are 1-3 cm depending on the country. Most patients with primary CMM > 4 mm are operated on with a margin of 2-cm today. The different national guidelines are thus, somewhat confusing and in a report from 2004 Thomas JM et al. showed that a 1-cm margin for CMM with a poor prognosis (≥2 mm) is associated with a greater risk of regional recurrence than in a 3-cm margin, but with a similar survival rate.

Today, according to Sladden et al. (2018), there have been published six randomized controlled trials (RCTs) assessing outcomes for surgical excision margins based upon Breslow thickness of invasive tumors. Three out of those six RCTs have included patients with CMMs 2-4 cm thick. Still, there are controversies and this report points out gaps of knowledge, e.g. lack of evidence about the optimal depth of excision and the optimal and minimal excision margins, since 1-cm versus 2-cm resection margins of invasive CMMs have not been directly compared yet.

Interestingly, out of one of the three RCTs analyzing melanomas with 2-4 mm thickness, long-term follow up data has recently been published by Hayes et al. 2016. They report an extended follow-up with a median follow-up of almost 9 years, concluding that 1-cm margin is not safe for high-risk CMMs compared to 3-cm margin.

From this point, based up on those interesting results, the investigators now present long-term follow-up of survival in patients included in the RCT published 2011 by Gillgren et al.

The original trial by Gillgren et al. 2011, is a randomized multicenter trial, launched from the Swedish Melanoma Study Group and the Danish Melanoma Group in 1992, included 936 patients from January 22 1992 to May 19 2004. Patients were recruited from Sweden (6 centers with 644 pat), Denmark (180 pat), Estonia (80 pat) and Norway (32 pat). Randomization routines were set up by the steering committee and eligible patients were randomized locally by telephone calls to national and international cancer centers (upon a histologically proven diagnoses and signed patient consent form). Only patients with a CMM >2 mm and with localized disease (who fulfilled the in- and exclusion criteria) were eligible for study inclusion. Patients with CMM on the hands, feet, head-neck and ano-genital region were excluded. Final surgery must had been planned within 8 weeks after date of diagnosis. All analyses were conducted according to the intention-to-treat principle.

Patients were followed clinically every 3 months for 2 years and thereafter every 6 months up to 5 years, with a median follow-up of 6.7 years. Follow-up data was thus collected from cancer registries, cause of death registries and medical records.

Statistical analyses were made by Kaplan Meier life-table curves. Prognostic factors were assessed with the use of a uni- and multivariate Cox regression analysis.

In the original study, the primary melanomas were removed either by an excisional biopsy (margin of 1-3 mm) or with a 2-cm margin before randomization. Patients were randomly assigned (1:1) to either a 2-cm surgical excision margin or a 4-cm surgical excision margin. The physician enrolled the patients after histological confirmation of melanomas >2 mm. Patients who had a diagnostic initial excision were randomized to the 2-cm group or to an additional wide local excision with a margin of up to either 2 cm or 4 cm. Patients who had a 2 cm initial excision were allocated to either no further surgery and randomized to the 2-cm group. Radical surgery was to be performed within 8 weeks after the date of diagnosis. The method of surgery was to extend to, or include, the deep fascia. Pathological excision margins were not registered. The sentinel node biopsy technique was introduced in the end of the enrolment period and was allocated to the same follow-up as the other patients. There were no protocol violations since the sentinel node biopsies were all in clinical stage IIA-C preoperatively. The patients were followed by standard clinical routines within participating centers at that time every 3 months for 2 years and then every 6 months until 5 years. Data on clinical relapse were obtained at the follow-up visits. Outcome data were also assessed from regional cancer registries, the national cause-of-death registries, and medical records.

In the long-term follow-up study, each country collected date of death, primary cause of death and underlying cause of death from central registries. The entire cohort was followed-up until Dec 31, 2016.

ELIGIBILITY:
Inclusion Criteria:

* Melanoma >2 mm
* Age ≤ 75 yr
* Patients operated on with ≤ 2-cm at diagnosis
* Final surgery planned within 8 weeks after date of diagnosis
* Patient fit for surgery
* Signed patient consent form

Exclusion Criteria:

* Melanoma on hand, foot, head-neck or ano-genital regions
* The presence of in-transit- regional and/or distant spread of the disease
* Illness making patient unfit for surgery
* Previous malignancies except basal cell- and in-situ colli uteri cancer

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 936 (Actual)
Dates: Start 1992-01; Primary Completion 2004-05 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Melanoma-specific survival | 24.9 years
  Cause of death: cutaneous malignant melanoma

SECONDARY OUTCOMES:
Overall survival | 24.9 years
  Cause of death: all death causes

CONTACTS AND LOCATIONS:
Overall Officials: Ulrik Ringborg, M.D., Ph.d., Principal Investigator — Karolinska inteitutet

IPD SHARING:
Plan to Share IPD: Undecided
Data could be shared with other researchers in a worldwide meta analysis after the actual study is completed.

REFERENCES:
- [Background] Gillgren P, Drzewiecki KT, Niin M, Gullestad HP, Hellborg H, Mansson-Brahme E, Ingvar C, Ringborg U. 2-cm versus 4-cm surgical excision margins for primary cutaneous melanoma thicker than 2 mm: a randomised, multicentre trial. Lancet. 2011 Nov 5;378(9803):1635-42. doi: 10.1016/S0140-6736(11)61546-8. Epub 2011 Oct 23. PMID 22027547
- [Background] Thomas JM, Newton-Bishop J, A'Hern R, Coombes G, Timmons M, Evans J, Cook M, Theaker J, Fallowfield M, O'Neill T, Ruka W, Bliss JM; United Kingdom Melanoma Study Group; British Association of Plastic Surgeons; Scottish Cancer Therapy Network. Excision margins in high-risk malignant melanoma. N Engl J Med. 2004 Feb 19;350(8):757-66. doi: 10.1056/NEJMoa030681. PMID 14973217
- [Background] Hayes AJ, Maynard L, Coombes G, Newton-Bishop J, Timmons M, Cook M, Theaker J, Bliss JM, Thomas JM; UK Melanoma Study Group; British Association of Plastic; Reconstructive and Aesthetic Surgeons, and the Scottish Cancer Therapy Network. Wide versus narrow excision margins for high-risk, primary cutaneous melanomas: long-term follow-up of survival in a randomised trial. Lancet Oncol. 2016 Feb;17(2):184-192. doi: 10.1016/S1470-2045(15)00482-9. Epub 2016 Jan 12. PMID 26790922
- [Background] Ethun CG, Delman KA. The importance of surgical margins in melanoma. J Surg Oncol. 2016 Mar;113(3):339-45. doi: 10.1002/jso.24111. Epub 2015 Dec 10. PMID 26662509
- [Background] Sladden MJ, Nieweg OE, Howle J, Coventry BJ, Thompson JF. Updated evidence-based clinical practice guidelines for the diagnosis and management of melanoma: definitive excision margins for primary cutaneous melanoma. Med J Aust. 2018 Feb 19;208(3):137-142. doi: 10.5694/mja17.00278. PMID 29438650
- [Derived] Utjes D, Malmstedt J, Teras J, Drzewiecki K, Gullestad HP, Ingvar C, Eriksson H, Gillgren P. 2-cm versus 4-cm surgical excision margins for primary cutaneous melanoma thicker than 2 mm: long-term follow-up of a multicentre, randomised trial. Lancet. 2019 Aug 10;394(10197):471-477. doi: 10.1016/S0140-6736(19)31132-8. Epub 2019 Jul 4. PMID 31280965